CLINICAL TRIAL: NCT03458728
Title: A Non-randomized, Open-label, Multi-center, Phase I/II Study of Phosphatidylinositol-3-kinase (PI3K) Inhibitor Copanlisib in Pediatric Patients With Relapsed/Refractory Solid Tumors or Lymphoma
Brief Title: Safety, Tolerability, Efficacy and Pharmacokinetics of Copanlisib in Pediatric Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no anticipated benefit over available standard therapies
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19176; 2017-000383-15 (EudraCT Number)
Record Dates: First submitted 2018-02-19; First posted 2018-03-08 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Relapsed or Refractory Solid Tumors or Lymphoma in Children; Neuroblastoma; Osteosarcoma; Rhabdomyosarcoma; Ewing Sarcoma
Keywords: Phase I: relapsed or refractory solid tumors or lymphoma; Phase II: relapsed or refractory solid tumors (neuroblastoma, osteosarcoma, rhabdomyosarcoma or Ewing sarcoma)
MeSH Terms: conditions — Recurrence; Neuroblastoma; Osteosarcoma; Rhabdomyosarcoma; Sarcoma, Ewing; Lymphoma | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose escalation of BAY806946 in Phase 1 (Experimental): It is estimated that 2 or 3 dose cohorts may be evaluated in phase 1 of the study. Safety and MTD/RP2D dose will be evaluated in 2 age groups (< 1 year old and ≥ 1 year old).
  Interventions: Drug: Copanlisib (BAY806946)
- Patients with Neuroblastoma in Phase 2 (Experimental): Recommended Phase 2 dose (RP2D) for copanlisib in pediatric patients, as defined in the Phase I part of the study, will be used.
  Interventions: Drug: Copanlisib (BAY806946)
- Patients with Osteosarcoma in Phase 2 (Experimental): RP2D for copanlisib in pediatric patients, as defined in the Phase I part of the study, will be used.
  Interventions: Drug: Copanlisib (BAY806946)
- Patients with Rhabdomyosarcoma in Phase 2 (Experimental): RP2D for copanlisib in pediatric patients, as defined in the Phase I part of the study, will be used.
  Interventions: Drug: Copanlisib (BAY806946)
- Patients with Ewing sarcoma in Phase 2 (Experimental): RP2D for copanlisib in pediatric patients, as defined in the Phase I part of the study, will be used.
  Interventions: Drug: Copanlisib (BAY806946)

INTERVENTIONS:
Drug: Copanlisib (BAY806946) — Copanlisib will be dosed on Day 1, Day 8, and Day 15 of every 28-day cycle. Phase 1: 2 or 3 dose cohorts may be evaluated in phase 1 of the study. Phase 2: RP2D for copanlisib in pediatric patients, as defined in the Phase I part of the study, will be used.

SUMMARY:
This study is designed to investigate whether the use of copanlisib is safe, feasible and beneficial to pediatric patients with solid solid tumors or lymphoma that are recurrent or refractory to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form by patients and/or patients' parents/legal guardians and age appropriate assent form by the patients obtained before any study specific procedure
* Male or female patients from 6 months to ≤ 21 years old at the time of study enrollment
* Confirmation of diagnosis:

  * Phase I: Patients must have histologic verification of a solid tumor or lymphoma malignancy at diagnosis, with measurable or evaluable disease, for which there is no standard curative anti-cancer treatment or treatment is no longer effective and must have received ≥ 1 prior line of therapy.
  * Phase II: patients must have histologically verified tumor at initial diagnosis and radiologically or histologically confirmed status at inclusion as indicated in the following: neuroblastoma, osteosarcoma, rhabdomyosarcoma or Ewing sarcoma.
  * Patients with solid tumors must have measurable disease (evaluable disease is acceptable for neuroblastoma and Ewing sarcoma). Tumor assessment will be done via computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography-computed tomography (PET-CT). Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, may be considered measurable if there has been demonstrated progression in the lesion. Bone scans (if clinically indicated) should be obtained within ≤ 4 weeks prior to the start of treatment.
* Performance level: Lansky ≥ 50% for patients ≤ 16 years of age and Karnofsky ≥ 50% for patients > 16 years of age.
* Adequate bone marrow, renal and liver function.

Exclusion Criteria:

* Active or uncontrolled infection (National Cancer Institute (NCI)-CTCAE Grade ≥ 2).
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator).
* Diabetes mellitus.
* Uncontrolled arterial hypertension despite optimal medical management (per institutional guidelines).
* Patients with central nervous system (CNS) malignancies.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - The Children's Hospital, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital For Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/19176
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 centers in United States between 30 APR 2018 (First participant first visit) and 1-Feb-2023 (Last participant last visit).
Pre-assignment Details: 41 participants were screened into the study (signed informed consent form (ICF)). 10 participants were screening failed. 31 participants were enrolled in the study, all 31 participants received treatment in phase 1 as the study was terminated prior to the initiation of the phase 2.
Groups:
- Copanlisib 28mg/m*2, Total: Copanlisib was administered Intravenous (IV) on Days 1, 8 and 15 of each 28-day treatment cycle. Treatment was continued until radiological progressive disease, unacceptable toxicity, withdrawal of consent, death or other event specified by the protocol. Copanlisib 28mg/m*2 (Total) included AMD0 (5 participants who were under the original DLT criteria) and AMD1+ (19 participants who were under the amended DLT criteria).
- Copanlisib 35mg/m*2: Copanlisib was administered Intravenous (IV) on Days 1, 8 and 15 of each 28-day treatment cycle. Treatment was continued until radiological progressive disease, unacceptable toxicity, withdrawal of consent, death or other event specified by the protocol.
Period: Overall Study
Arm/Group | Copanlisib 28mg/m*2, Total | Copanlisib 35mg/m*2
Started | 24 | 7
Started Treatment | 24 | 7
Terminated Treatment | 24 | 7
Completed | 0 | 0
Not Completed | 24 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Progressive disease - clinical assessment | 1 | 0
Not completed — Progressive disease - radiological progression | 21 | 6
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Copanlisib 28mg/m*2, Total | Copanlisib 35mg/m*2 | Total
Number analyzed (Participants) | 24 | 7 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (4.6) | 12.3 (3.8) | 12.5 (4.3)
Age, Customized [Number; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 11 | 3 | 14
  Adolescents (12-17 years) | 10 | 4 | 14
  Adults (18-64 years) | 3 | 0 | 3
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 14 | 4 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 18 | 6 | 24
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 17 | 3 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: The Maximum Tolerated Dose (MTD): the Highest Dose Level of Copanlisib That Can be Given so That Not More Than 1 Out of 6 Patients Experience a DLT During the DLT Evaluation Period.
Description: Maximum tolerated dose (MTD) for copanlisib was defined as the highest dose level where 6 patients have been treated and ≤ 1 participant experienced a DLT. This endpoint was performed on SAF.
Time Frame: Cycle 1 (28 days)
Population: Safety analysis set (SAF): The SAF population was defined as all participants with at least one intake of study drug.
Measure: Number; unit: mg/m*2/dose
Groups:
- Copanlisib_Phase 1: Copanlisib was administered on Day 1, Day 8, and Day 15 of every 28-day cycle. Subjects received copanlisib IV infusion with intermittent (3 weeks on / 1 week off) dosing schedule at the assigned dose level.
Arm/Group | Copanlisib_Phase 1
Number analyzed (Participants) | 31
mg/m*2/dose | 28

2. Primary Outcome: Phase 1: Number of Subjects With Dose Limiting Toxicity (DLT)
Description: DLT was observed during first cycle of treatment, and assessed as possibly, probably or definitely related to treatment with copanlisib. The DLT observation period for the purposes of dose-escalation was the first cycle of therapy.
Time Frame: Cycle 1 (28 days)
Population: Safety analysis set (SAF): The SAF population was defined as all participants with at least one intake of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Copanlisib 28mg/m*2, Total | Copanlisib 35mg/m*2
Number analyzed (Participants) | 24 | 7
Participants | 3 | 2

3. Primary Outcome: Phase 1: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: TEAE was defined as any event arising or worsening after start of study drug administration until 30 days after the last dose of the study drug intake (end of safety follow-up).
  This endpoint was performed on SAF.
Time Frame: After the first study intervention up to 30 days after the last dose of the study drug intake (end of safety follow up), with a maximum of 145 days.
Population: Safety analysis set (SAF): The SAF population was defined as all participants with at least one intake of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Copanlisib 28mg/m*2, Total | Copanlisib 35mg/m*2
Number analyzed (Participants) | 24 | 7
Participants | 24 | 7

4. Primary Outcome: Phase 1: Number of Subjects With Serious Adverse Events (SAEs)
Description: This endpoint was performed on SAF.
Time Frame: Up to 150 days.
Population: Safety analysis set (SAF): The SAF population was defined as all participants with at least one intake of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Copanlisib 28mg/m*2, Total | Copanlisib 35mg/m*2
Number analyzed (Participants) | 24 | 7
Participants | 10 | 0

5. Primary Outcome: Phase 1: Number of Participants With Treatment-related Adverse Events (AEs).
Description: This endpoint was performed on SAF.
Time Frame: Up to 145 days.
Population: Safety analysis set (SAF): The SAF population was defined as all participants with at least one intake of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Copanlisib 28mg/m*2, Total | Copanlisib 35mg/m*2
Number analyzed (Participants) | 24 | 7
Participants | 5 | 0

6. Primary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR was defined separately in each indication, as the number of responders divided by the number of subjects in FAS in the indication.
Time Frame: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Population: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Groups:
- Copanlisib_Phase 2: As the study was terminated before the initiation of phase 2, data was not collected in phase 2.
Arm/Group | Copanlisib_Phase 2
Number analyzed (Participants) | 0

7. Primary Outcome: Phase 2: Disease Control Rate (DCR)
Description: The DCR was defined as the number of subjects with disease control divided by the number of subjects in FAS or per protocol set (PPS) in the indication.
Time Frame: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Population: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Arm/Group | Copanlisib_Phase 2
Number analyzed (Participants) | 0

8. Primary Outcome: Phase 2: Progression-free Survival (PFS)
Time Frame: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Population: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Arm/Group | Copanlisib_Phase 2
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase 1: Copanlisib Maximum Drug Concentration (Cmax)
Description: Cmax: maximum concentration after the 3rd dose in a sequence of 3 nominal doses of copanlisib.
  PK analysis set: All participants with at least one intake of study drug and with at least one valid measurement for copanlisib were included in the copanlisib PK analysis.
Time Frame: Age ≥ 6 years: Pre-dose, Post-dose on Cycle 1 Day 1 and Day 15 (1-1.25 hour (h), 1.5- 3h, 22-24h). Age < 6 years: Pre-dose, Post-dose on Cycle 1 Day 1 and Day 15 (1-1.25h, 22-24h). Cycle length is 28 days.
Population: For all participants included in the PK analysis set, copanlisib PK was analyzed using an established comprehensive population PK model with incorporation of allometric scaling by Body surface area (BSA) on copanlisib disposition parameters (clearance and volume parameters). The model with allometric scaling enables combining of treatment groups and was used to estimate copanlisib PK parameters (AUC0-168h and Cmax).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Copanlisib_Phase 1
Number analyzed (Participants) | 30
μg/L | 359 (22.6)

10. Secondary Outcome: Phase 1: Area Under the Curve (AUC(0-168))
Description: AUC(0-168): Area under the concentration-time curve [AUC] from 0 to 168 hours after the 3rd dose in a sequence of 3 nominal doses of copanlisib.
  PK analysis set: All participants with at least one intake of study drug and with at least one valid measurement for copanlisib were included in the copanlisib PK analysis.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg∙h/L
Arm/Group | Copanlisib_Phase 1
Number analyzed (Participants) | 30
μg∙h/L | 2900 (35.4)

11. Secondary Outcome: Phase 1: Objective Response Rate (ORR)
Description: ORR by dose cohort is defined as the number of responders divided by the number of subjects in FAS in the indication.
  The analysis of ORR was performed on FAS.
Time Frame: Up to 150 days
Population: Full analysis set (FAS): All subjects with at least one intake of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Copanlisib 28mg/m*2, Total | Copanlisib 35mg/m*2
Number analyzed (Participants) | 24 | 7
Participants | 0 | 0

12. Secondary Outcome: Phase 2: Duration of Response (DOR)
Time Frame: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Population: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Arm/Group | Copanlisib_Phase 2
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 2: PFS in Each Indication Except for Osteosarcoma
Time Frame: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Population: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Arm/Group | Copanlisib_Phase 2
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase 2: Overall Survival (OS)
Time Frame: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Population: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Arm/Group | Copanlisib_Phase 2
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 2: Number of Participants With Treatment-emergent AEs
Time Frame: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Population: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Arm/Group | Copanlisib_Phase 2
Number analyzed (Participants) | 0

16. Secondary Outcome: Phase 2: Number of Subjects With Treatment Emergent SAEs
Time Frame: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Population: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Arm/Group | Copanlisib_Phase 2
Number analyzed (Participants) | 0

17. Secondary Outcome: Phase 2: Number of Subjects With Treatment-emergent Clinically Significant Change in Laboratory Parameters, ECGs and Vital Signs
Time Frame: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Population: Data was not collected for this endpoint due to study was terminated before the initiation of phase 2.
Arm/Group | Copanlisib_Phase 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: After the first study intervention up to 30 days after the last dose of the study drug intake (end of safety follow up), with a maximum of 150 days. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, with a maximum of 150 days.
Groups:
- Copanlisib 35mg/m*2: Copanlisib was administered Intravenous (IV) on Days 1, 8 and 15 of each 28-day treatment cycle. Treatment was continued until radiological progressive disease,unacceptable toxicity, withdrawal of consent, death or other event specified by the protocol.
Arm/Group | Copanlisib 28mg/m*2, Total | Copanlisib 35mg/m*2
All-Cause Mortality (participants affected / at risk) | 20/24 | 5/7
Serious Adverse Events (participants affected / at risk) | 10/24 | 0/7
Other Adverse Events (participants affected / at risk) | 23/24 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copanlisib 28mg/m*2, Total (N=24) | Copanlisib 35mg/m*2 (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (8) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copanlisib 28mg/m*2, Total (N=24) | Copanlisib 35mg/m*2 (N=7)
Anaemia (Blood and lymphatic system disorders) | 13 (38) | 3 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (21) | 3 (4)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 6 (7) | 3 (4)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (9) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (6) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 2 (3)
Nausea (Gastrointestinal disorders) | 15 (22) | 4 (7)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (11) | 4 (12)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 10 (14) | 3 (7)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (19) | 4 (7)
Non-cardiac chest pain (General disorders) | 4 (5) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 6 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (8) | 1 (2)
Amylase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (11) | 2 (2)
Blood cholesterol increased (Investigations) | 5 (5) | 1 (1)
Blood creatinine increased (Investigations) | 4 (4) | 2 (4)
Blood lactate dehydrogenase increased (Investigations) | 5 (6) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0)
Carbon dioxide decreased (Investigations) | 3 (8) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
High density lipoprotein decreased (Investigations) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 3 (3) | 0 (0)
Lipase increased (Investigations) | 5 (7) | 0 (0)
Lymphocyte count decreased (Investigations) | 13 (35) | 3 (7)
Neutrophil count decreased (Investigations) | 6 (14) | 2 (9)
Neutrophil count increased (Investigations) | 2 (3) | 0 (0)
Protein total decreased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 3 (6) | 2 (3)
White blood cell count decreased (Investigations) | 12 (21) | 5 (7)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (44) | 4 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 6 (7) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (16) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (12) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (10) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (8) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (16) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (11) | 1 (1)
Hypouricaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (8) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (12) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (12) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 9 (11) | 1 (3)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Irritability (Psychiatric disorders) | 2 (3) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 10 (42) | 2 (2)
Hypotension (Vascular disorders) | 7 (7) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT03458728/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT03458728/SAP_001.pdf